CLINICAL TRIAL: NCT02011386
Title: Improved Monitoring and Prediction of Clinical Response and Disease Course During Golimumab Therapy of Patients With Axial Spondyloarthritis
Brief Title: Novel MRI ANd Biomarkers in GOlimumab-treated Patients With Axial Spondyloarthritis
Acronym: MANGO
Status: Completed | Type: Observational
Sponsor: Professor Mikkel Østergaard (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Professor Mikkel Østergaard, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: MANGO
Record Dates: First submitted 2013-12-06; First posted 2013-12-13 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment: Treatment: Injection Golimumab 50 mg every month on the same date
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment
  Other Names: Treatment: Injection Golimumab 50 mg every month on the same date

SUMMARY:
The study investigates different criteria for remission based on MRI and circulating biomarkers for inflammation, cartilage, connective tissue and bone turnover in patients with axial spondyloarthritis treated with Golimumab. Furthermore, the study also investigates factors that affect disease activity, function and participation by use of different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Axial spondyloarthritis according to the Assessment of Spondyloarthritis International Society (ASAS) classification criteria for axial spondyloarthritis
* Sacroiliitis on conventional X-rays or Magnetic Resonance Imaging (MRI).
* Disease activity assessed by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >40 mm despite treatment with Non-Steroidal Anti-Inflammatory Drugs (NSAID).
* Clinical indication for tumor necrosis factor (TNF) inhibitor treatment by the treating physician.

Exclusion Criteria:

* No contraindications for TNF inhibitor
* No contraindications for MRI
* No contraindications in participation in a study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with axial spondyloarthritis with moderate to high disease activity (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at least 40 mm), who are going to start treatment with TNF inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, Professor, Principal Investigator — Glostrup Hospital, University of Copenhagen
Locations (6):
- Denmark (6):
  - Frederiksberg Bispebjerg Hospitals, Dep. of Rheumatology, Copenhagen
  - Glostrup Hospital, Dep. of Rheumatology, Copenhagen
  - Herlev Hospital, Dep. of Radiology, Copenhagen
  - Gentofte Hospital, Dep. of Rheumatology, Copenhagen
  - Nordsjællands Hospital Hillerød, Dep. of Rheumatology, Hillerød
  - Køge Hospital, Dep. of Rheumatology, Køge

REFERENCES:
- [Derived] Lorincz M, Ostergaard M, Wetterslev M, Sorensen IJ, Madsen OR, Christiansen SN, Hetland ML, Bakkegaard M, Klarlund M, Duer A, Boesen M, Gosvig KK, Pedersen SJ. Construct validity and responsiveness of ASAS Health Index assessed in two longitudinal studies of tumour necrosis factor alpha inhibitor initiation and dose reduction in patients with axial spondyloarthritis. RMD Open. 2024 Dec 20;10(4):e004948. doi: 10.1136/rmdopen-2024-004948. PMID 39794273
- [Derived] Krabbe S, Eshed I, Sorensen IJ, Moller J, Jensen B, Madsen OR, Klarlund M, Pedersen SJ, Ostergaard M. Novel whole-body magnetic resonance imaging response and remission criteria document diminished inflammation during golimumab treatment in axial spondyloarthritis. Rheumatology (Oxford). 2020 Nov 1;59(11):3358-3368. doi: 10.1093/rheumatology/keaa153. PMID 32310294
- [Derived] Krabbe S, Ostergaard M, Pedersen SJ, Weber U, Krober G, Makysmowych W, Lambert RGW. Canada-Denmark MRI scoring system of the spine in patients with axial spondyloarthritis: updated definitions, scoring rules and inter-reader reliability in a multiple reader setting. RMD Open. 2019 Oct 13;5(2):e001057. doi: 10.1136/rmdopen-2019-001057. eCollection 2019. PMID 31673422

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 53
Completed | 48
Not Completed | 5
Not completed — Non-compliance | 2
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [28 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 53
Fulfilment of the radiographic part of the modified New York criteria [Count of Participants; unit: Participants] — Each sacroiliac joint is assigned a score of 0 to 4 based on the appearance on a radiograph, grade 0 is normal, grade 1 is suspicious changes, grade 2 is minimum abnormality, grade 3 is unequivocal abnormality and grade 4 is severe abnormality. A patient fulfils the radiographic part of the modified New York criteria if there is sacroiliitis of at least grade 2 bilaterally or sacroiliitis grade 3 or 4 unilaterally. Reference: Arthritis Rheum 1984;27:361-8.
  Participants | 33
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 24 [21 to 28]
Symptom duration [Median (Inter-Quartile Range); unit: years] | 5.1 [2.6 to 12.8]
Positive for HLA-B27 [Count of Participants; unit: Participants] | 40
hsCRP [Median (Inter-Quartile Range); unit: mg/L] — C-reactive protein. The assay had a lower limit of detection of 0.3 mg/L.
  mg/L | 6.8 [1.3 to 19]
Ankylosing Spondylitis Disease Activity Score (ASDAS) [Median (Inter-Quartile Range); unit: units on a scale] — ASDAS is a composite index to assess disease activity in axSpA. ASDAS parameters: 1) Total back pain 2) Patient global 3) Peripheral pain/swelling 4) Duration of morning stiffness 5) CRP in mg/L: ASDAS calculation: 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(max(CRP,2)+1). CRP is in milligram/liter (mg/L), the range of other variables is from 0 to 10. Data from five variables combine to yield a score (minimum 0.636 to no defined upper limit), higher scores indicate higher disease activity.
  units on a scale | 3.6 [3.1 to 4.1]
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Median (Inter-Quartile Range); unit: units on a scale] — BASDAI is a measure of disease activity which was calculated based on 6 separate questionnaire items that were answered by the patients using visual analogue scale scales with range 0-10. A weighted average was performed, where items 5 and 6 had a weight of 0.5 whereas items 1, 2, 3 and 4 had a weight of 1. Range is from 0 to 10, with 10 indicating more severe disease activity.
  units on a scale | 6.2 [5.1 to 7.1]
Bath Ankylosing Spondylitis Functional Index (BASFI) [Median (Inter-Quartile Range); unit: units on a scale] — BASFI is a measure of physical function which was calculated based on 10 separate questionnaire items that were answered by the patients using visual analogue scales with range 0-10, an average across 10 items was calculated. The range is 0-10 with 10 indicating that the level of physical functioning is more severely affected.
  units on a scale | 4.6 [3.2 to 6.1]
Bath Ankylosing Spondylitis Metrology Index (BASMI) [Median (Inter-Quartile Range); unit: units on a scale] — 5 components of BASMI were each scored 0, 1 or 2, based on physical examination tests of the range of motion of the vertebral column and hips. The scores were added, and the range was 0-10, where 10 indicates a worse metrology (i.e. more severely affected range of motion of the vertebral column and hips).
  units on a scale | 2 [1 to 3]
Chest expansion [Median (Inter-Quartile Range); unit: cm] | 4.0 [3.0 to 5.0]
Swollen joint count of 66 joints [Median (Inter-Quartile Range); unit: joints] | 0 [0 to 0]
Tender joint count of 68 joints [Median (Inter-Quartile Range); unit: joints] | 0 [0 to 3]
Tender enthesis count [Median (Inter-Quartile Range); unit: entheses] — Range is 0-35. The entheses assessed were those that are included in either the Maastricht Ankylosing Spondylitis Enthesitis Score (MASES), the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis index or the Leeds Enthesitis Index (LEI).
  entheses | 3 [2 to 6]
Pain score [Median (Inter-Quartile Range); unit: units on a scale] — Questionnaire filled in by the patient, visual analogue scale with range 0-10, 10 indicates more severe pain.
  units on a scale | 6.9 [5.5 to 8.0]
Patient's global score [Median (Inter-Quartile Range); unit: units on a scale] — Questionnaire filled in by the patient to capture the global disease activity as assessed by the patient; visual analogue scale with range 0-10, 10 indicates worse global score
  units on a scale | 7.5 [6.5 to 8.4]
Physician's global score [Median (Inter-Quartile Range); unit: units on a scale] — Questionnaire filled in by the physician to capture the physician's global assessment of disease activity; visual analogue scale with range 0-10, 10 indicates a worse disease activity.
  units on a scale | 4.9 [3.3 to 6.4]
Modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) [Median (Inter-Quartile Range); unit: units on a scale] — The mSASSS is an assessment of structural lesions of the spine using lateral radiographs of the cervical and lumbar spine. The mSASSS is the sum of the lumbar and cervical spine score (range 0 [no change] to 72 [severe change]), derived from scoring the anterior sites of the lumbar spine (T12 to S1) and the cervical spine (C2 to T1) as either 0 (normal), 1 (erosion, sclerosis, or squaring), 2 (syndesmophyte), 3 (bridging syndesmophyte), and adding all scores together.
  units on a scale | 0 [0 to 1]
Canada-Denmark (CANDEN) Magnetic Resonance Imaging (MRI) Spine Inflammation Index [Median (Inter-Quartile Range); unit: units on a scale] — Semiquantitative score of inflammation of the spine as assessed by MRI. A comprehensive assessment system is applied to different anatomical parts of the spine at 23 spinal levels and all scores are summed; range is 0-614 with higher scores indicating more severe inflammation. Reference: RMD Open 2019;5:e001057.
  units on a scale | 8 [2 to 16]
Canada-Denmark (CANDEN) Magnetic Resonance Imaging (MRI) Spine Fat Metaplasia Score [Median (Inter-Quartile Range); unit: units on a scale] — Semiquantitative score of fat metaplasia of the spine as assessed by MRI. A comprehensive assessment system is applied to different anatomical parts of the spine at 23 spinal levels and all scores are summed; range is 0-510 with higher scores indicating more severe fat metaplasia. Reference: RMD Open 2019;5:e001057.
  units on a scale | 3 [0 to 13]
Canada-Denmark (CANDEN) Magnetic Resonance Imaging (MRI) Spine Erosion Score [Median (Inter-Quartile Range); unit: units on a scale] — Semiquantitative score of erosion of the spine as assessed by MRI. A comprehensive assessment system is applied to different anatomical parts of the spine at 23 spinal levels and all scores are summed; range is 0-208 with higher scores indicating more severe erosion. Reference: RMD Open 2019;5:e001057.
  units on a scale | 0 [0 to 0]
Canada-Denmark (CANDEN) Magnetic Resonance Imaging (MRI) Spine New Bone Formation Score [Median (Inter-Quartile Range); unit: units on a scale] — Semiquantitative score of new bone formation of the spine as assessed by MRI. A comprehensive assessment system is applied to different anatomical parts of the spine at 23 spinal levels and all scores are summed; range is 0-460 with higher scores indicating more severe new bone formation. Reference: RMD Open 2019;5:e001057.
  units on a scale | 0 [0 to 8]
SPARCC MRI Spine Inflammation Index [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Spine Inflammation Index. 23 levels of the spine are assessed for the presence, intensity and depth of inflammation at a maximum of 3 slices per level, and scores are summed together. Range is 0-414 with higher scores indicating more severe inflammation of the spine.
  units on a scale | 8 [4 to 16]
SPARCC MRI Sacroiliac Joint Inflammation Index [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac Joint Inflammation Index as based on an assessment of the presence, depth and intensity of inflammation as assessed on 6 MRI slices, and all scores are summed together; range is 0-72, with higher scores indicating more severe inflammation of the sacroiliac joints.
  units on a scale | 13 [3 to 22]
SPARCC MRI Sacroiliac Joint Structural Score - Fat [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac Joint Structural Score - Fat is based on an assessment of MRI images of the sacroilliac joints where the presence of fat is assessed on 5 MRI slices; range is 0-40, with higher scores indicating worse fat metaplasia.
  units on a scale | 2 [0 to 12]
SPARCC MRI Sacroiliac Joint Structural Score - Erosion [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac Joint Structural Score - Erosion is based on an assessment of MRI images of the sacroilliac joints where the presence of erosion is assessed on 5 MRI slices; range is 0-40, with higher scores indicating worse erosion.
  units on a scale | 6 [1 to 10]
SPARCC MRI Sacroiliac Joint Structural Score - Backfill [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac Joint Structural Score - Backfill is based on an assessment of MRI images of the sacroilliac joints where the presence of backfill is assessed on 5 MRI slices; range is 0-20, with higher scores indicating worse backfill. According to the recently updated terminology by Assessment of Spondyloarthritis International Society MRI Group, backfill is termed "fat metaplasia in an erosion cavity".
  units on a scale | 0 [0 to 2]
SPARCC MRI Sacroiliac Joint Structural Score - Ankylosis [Median (Inter-Quartile Range); unit: units on a scale] — Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac Joint Structural Score - Ankylosis is based on an assessment of MRI images of the sacroilliac joints where the presence of ankylosis is assessed on 5 MRI slices; range is 0-20, with higher scores indicating worse ankylosis.
  units on a scale | 0 [0 to 0]
MRI Peripheral Joints and Entheses Inflammation Index [Median (Inter-Quartile Range); unit: units on a scale] — Magnetic Resonance Imaging (MRI) Peripheral Joints and Entheses Inflammation Index was based on an assessment of MRI images of several image stations: anterior chest wall and shoulder, hands, pelvis, knees, ankles and feet; 74 joints were assessed for synovitis and osteitis, 30 entheses were assessed for soft tissue inflammation and osteitis, and all scores were summed together; range was 0-210, with higher scores indicating worse inflammation of joints and entheses throughout the body as assessed by MRI.
  units on a scale | 7 [4 to 14]
Assessment of Spondyloarthritis International Society (ASAS) criteria: Inflammatory back pain [Count of Participants; unit: Participants] — IBP according to experts: four out of five of the following parameters present: (1) age at onset less than 40 years, (2) insidious onset, (3) improvement with exercise, (4) no improvement with rest, (5) pain at night (with improvement upon getting up). (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 50
Assessment of Spondyloarthritis International Society (ASAS) criteria: Arthritis [Count of Participants; unit: Participants] — Past or present active synovitis diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 12
Assessment of Spondyloarthritis International Society (ASAS) criteria: Heel enthesitis [Count of Participants; unit: Participants] — Heel enthesitis: past or present spontaneous pain or tenderness at examination at the site of the insertion of the Achilles tendon or plantar fascia at the calcaneus. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 12
Assessment of Spondyloarthritis International Society (ASAS) criteria: Uveitis [Count of Participants; unit: Participants] — Past or present uveitis anterior, confirmed by an ophthalmologist. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 9
Assessment of Spondyloarthritis International Society (ASAS) criteria: Dactylitis [Count of Participants; unit: Participants] — Past or present dactylitis diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 3
Assessment of Spondyloarthritis International Society (ASAS) criteria: Psoriasis [Count of Participants; unit: Participants] — Past or present psoriasis diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 6
Assessment of Spondyloarthritis International Society (ASAS) criteria: Inflammatory bowel disease [Count of Participants; unit: Participants] — Past or present Crohn disease or ulcerative colitis diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 2
Assessment of Spondyloarthritis International Society (ASAS) criteria: Good response to NSAIDs [Count of Participants; unit: Participants] — At 24-48 h after a full dose of NSAID the back pain is not present anymore or much better. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 38
Assessment of Spondyloarthritis International Society criteria: Family history of spondyloarthritis [Count of Participants; unit: Participants] — Presence in first-degree or second-degree relatives of any of the following: (a) ankylosing spondylitis, (b) psoriasis, (c) uveitis, (d) reactive arthritis, (e) inflammatory bowel disease. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 15
Assessment of Spondyloarthritis International Society (ASAS) criteria: Elevated C-reactive protein [Count of Participants; unit: Participants] — CRP above upper normal limit in the presence of back pain, after exclusion of other causes for elevated CRP concentration. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 34
csDMARDs at baseline [Count of Participants; unit: Participants] — Conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) were allowed, but the dose could not be changed 4 weeks prior to baseline.
  Participants
    Sulfasalazine at baseline | 2
    Methotrexate at baseline | 1
    Leflunomide at baseline | 1
    No csDMARDs | 49

OUTCOME MEASURES:

1. Primary Outcome: Fulfillment of Bath Ankylosing Spondylitis Disease Activity Index 50 Response (BASDAI50)
Description: At least 50% reduction in BASDAI score at follow-up compared with BASDAI score at baseline
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 31

2. Secondary Outcome: BASDAI 50% or 2.0 Improvement
Description: At least 50% decrease or at least an improvement of 2.0 in BASDAI, when measured on a scale with range 0-10.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 36

3. Secondary Outcome: BASDAI 50% or 2.0 Improvement
Description: At least 50% decrease or at least an improvement of 2.0 in BASDAI, when measured on a scale with range 0-10.
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 36

4. Secondary Outcome: Ankylosing Spondylitis Disease Activity Score Clinically Important Improvement (ASDAS-CII)
Description: Decrease in ASDAS score at follow-up compared with ASDAS score at baseline of at least 1.1.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 40

5. Secondary Outcome: Ankylosing Spondylitis Disease Activity Score Clinically Important Improvement (ASDAS-CII)
Description: Decrease in ASDAS score at follow-up compared with ASDAS score at baseline of at least 1.1.
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 34

6. Secondary Outcome: MRI Spine Remission
Description: Maximum 1 disco-vertebral unit with inflammation present.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 32

7. Secondary Outcome: MRI-SPINE-50
Description: At least 50% reduction in Canada-Denmark (CANDEN) MRI spine inflammation score.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 30

8. Other Pre Specified Outcome: MRI-SIJ-50
Description: At least 50% decrease in Spondyloarthritis Research Consortium of Canada (SPARCC) MRI sacroiliac joint inflammation index
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 29

9. Other Pre Specified Outcome: MRI-PERIPH-50
Description: At least 50% reduction in MRI Peripheral Joints and Entheses Inflammation Index. MRIs of 74 peripheral joints were evaluated separately for synovitis and osteitis (i.e. bone marrow edema) and 30 peripheral entheses were evaluated separately for soft tissue inflammation and osteitis. All types of lesions (i.e. joint synovitis, joint osteitis, entheseal soft tissue inflammation and entheseal osteitis) were scored on a semi-quantitative scale of 0-2 ('none', 'mild', 'moderate to severe').
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 17

10. Other Pre Specified Outcome: MRI SI Joint Remission
Description: Inflammation in 2 or fewer quadrants as assessed slice by slice across MRI slices that depict the cartilagenous compartment of the sacroiliac joints.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 24

11. Other Pre Specified Outcome: MRI Peripheral Joints and Entheses Inflammation Remission
Description: A score of maximally 2 of the MRI Peripheral Joints and Entheses Inflammation Index.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of start of golimumab treatment and until the date of the week 52 visit or the date of early termination.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 20/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=53)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (9)
Fatigue (General disorders) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT02011386/Prot_SAP_000.pdf